CLINICAL TRIAL: NCT03702322
Title: Improving Voice Production for Adults With Age-related Dysphonia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21DC016356 (NIH)
Record Dates: First submitted 2018-09-17; First posted 2018-10-11 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Presbylarynx; Age-Related Dysphonia

STUDY DESIGN:
Intervention Model Description: All participants receive every intervention in randomized order
Masking Description: Participants in the perceptual studies rating audio and visual files will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): All participants will undergo each treatment.
  Interventions: Behavioral: Voice therapy: respiratory; Behavioral: Voice therapy: glottal closure; Behavioral: Voice therapy: loud; Behavioral: Voice therapy: Semiocclusion

INTERVENTIONS:
Behavioral: Voice therapy: respiratory — Abdominal voice onset
Behavioral: Voice therapy: glottal closure — Pulling/pushing task
Behavioral: Voice therapy: loud — Assertive task
Behavioral: Voice therapy: Semiocclusion — Semi-occluded vocal tract

SUMMARY:
The objectives for this research are to determine the mechanisms by which specific therapy tasks improve voice in age-related dysphonia, and the conditions that limit the extent of improvement. The central hypothesis is that targeted therapy tasks will improve voice, and that severity will determine the extent of improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adults in age range who volunteer
* Can understand and complete directions presented in English
* People with voice disorder associated with advancing age will be included, including bowing, incomplete closure, mild edema, erythema, signs of laryngopharyngeal reflux.

Exclusion Criteria:

* Laryngeal differences not related to aging (e.g., vocal fold paralysis, moderate-severe edema, lesions, leukoplakia, dysplasia, Parkinson disease)
* Known history of stroke, brain injury, or other neurological disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Relative glottal gap from laryngeal high-speed videoendoscopy | End of year 3
Perceived voice quality | End of year 3
  Participants will score the construct of "overall voice quality" using a technique called "sort and rate" in which listeners move icons representing each sound along a line. They align the icons so that best voices are on one side and worst voices are on the other. The distance between the icons represents how much better or worse one sound is than the other. There are no units to the scale. Rankings from all listeners are combined using the statistical technique of multidimensional scaling. The result is a ranked value for each sound file (i.e., voice production) that shows how different they are. There is no highest or lowest value.
Acoustic measure of voice quality (Cepstral Peak Prominence) | End of year 3

SECONDARY OUTCOMES:
Open quotient from laryngeal high-speed videoendoscopy | End of year 3
Speed index from laryngeal high-speed videoendoscopy | End of year 3
Maximum area declination ratefrom laryngeal high-speed videoendoscopy | End of year 3
Fundamental frequency standard deviation from laryngeal high-speed videoendoscopy | End of year 3

CONTACTS AND LOCATIONS:
Overall Officials: Robin A Samlan, Ph.D., Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona